CLINICAL TRIAL: NCT01362894
Title: Clinical Comparison of Two Daily Disposable Toric Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-346-C-013
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-07

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nelfilcon A / etafilcon A (Other): Nelfilcon A lenses worn first, with etafilcon A lenses worn second. Both products worn bilaterally on a daily wear, daily disposable basis for one week each.
  Interventions: Device: nelfilcon A contact lens; Device: etafilcon A contact lens
- etafilcon A / nelfilcon A (Other): Etafilcon A lenses worn first, with nelfilcon A lenses worn second. Both products worn bilaterally on a daily wear, daily disposable basis for one week each.
  Interventions: Device: nelfilcon A contact lens; Device: etafilcon A contact lens

INTERVENTIONS:
Device: nelfilcon A contact lens — Commercially marketed, nelfilcon A, toric, soft contact lens for daily disposable wear.
  Other Names: Focus® DAILIES® Toric
Device: etafilcon A contact lens — Commercially marketed, etafilcon A, toric, soft contact lens for daily disposable wear.
  Other Names: 1-DAY ACUVUE® MOIST® FOR ASTIGMATISM

SUMMARY:
The purpose of this trial was to compare the performance of two contact lenses commercially available for people with astigmatism.

DETAILED DESCRIPTION:
This trial compared the performance of two commercialized daily disposable contact lenses in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent.
* Germany: Be of legal age.
* Current monthly or weekly toric soft lens wearer able to be fit in both eyes with soft toric lenses in the study parameters.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in an ophthalmic clinical trial.
* Wears contact lenses overnight while sleeping.
* Habitual daily disposable contact lens wearer.
* Monovision correction during the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled from 19 German study sites.
Pre-assignment Details: Two participants were enrolled, but not dispensed, due to unacceptable objective vision (1) and biomicroscopy findings (1). Baseline characteristics are presented on all enrolled and dispensed participants: 238.
Period: Period One, 1 Week
Arm/Group | Nelfilcon A / Etafilcon A | Etafilcon A / Nelfilcon A
Started | 119 (One participant was not dispensed lenses until Period 2.) | 117 (One participant was not dispensed lenses until Period 2.)
Completed | 119 | 117
Not Completed | 0 | 0
Period: Period Two, 1 Week
Arm/Group | Nelfilcon A / Etafilcon A | Etafilcon A / Nelfilcon A
Started | 118 (Two participants discontinued between Periods 1 and 2 due to discomfort (1) and poor fit (1).) | 115 (Three participants discontinued between Periods 1 and 2 due to unacceptable vision.)
Completed | 118 | 115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All enrolled and dispensed participants.
Arm/Group | Overall
Number analyzed (Participants) | 238
Age Continuous [Mean (Standard Deviation); unit: years] | 31.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159
  Male | 79
Region of Enrollment [Number; unit: participants]
  Germany | 238

OUTCOME MEASURES:

1. Primary Outcome: Overall Vision
Description: As interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 1 week of wear time. Overall vision was rated on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 1 week, replacing lenses daily
Population: The Efficacy Evaluable Set (EES) contained all enrolled and dispensed subjects with no major protocol deviations as determined by masked review that also completed a minimum of 4 days of lens wear with either study product and attended an assessing follow-up visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Nelfilcon A: Nelfilcon A lenses worn bilaterally on a daily wear, daily disposable basis for one week.
- Etafilcon A: Etafilcon A lenses worn bilaterally on a daily wear, daily disposable basis for one week.
Arm/Group | Nelfilcon A | Etafilcon A
Number analyzed (Participants) | 226 | 228
Units on a scale | 8.2 (1.7) | 7.5 (2.1)

2. Primary Outcome: Overall Comfort
Description: As interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 1 week of wear time. Overall comfort was rated on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 1 week, replacing lenses daily
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nelfilcon A | Etafilcon A
Number analyzed (Participants) | 227 | 229
Units on a scale | 7.8 (1.8) | 7.2 (2.0)

3. Primary Outcome: Overall Handling
Description: As interpreted by the participant and recorded on a questionnaire as a single, retrospective evaluation of 1 week of wear time. Overall handling was rated on a 10-point scale, with 1 being difficult and 10 being easy.
Time Frame: 1 week, replacing lenses daily
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nelfilcon A | Etafilcon A
Number analyzed (Participants) | 227 | 229
Units on a scale | 8.2 (1.8) | 6.8 (2.2)

4. Primary Outcome: Overall Satisfaction
Description: as for outcome 1
Time Frame: 1 week, replacing lenses daily
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nelfilcon A | Etafilcon A
Number analyzed (Participants) | 227 | 229
Units on a scale | 7.7 (1.9) | 6.9 (2.0)

5. Secondary Outcome: Ease of Selecting Final Lens Power
Description: As interpreted by the investigator at time of lens fitting and recorded on a questionnaire. Ease of selecting final lens power was rated on a 10-point scale, with 1 being difficult and 10 being easy.
Time Frame: Day 0
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nelfilcon A | Etafilcon A
Number analyzed (Participants) | 228 | 229
Units on a scale | 8.4 (1.5) | 8.8 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 20-May-2011 to 15-AUG-2011.
Description: The safety population included all enrolled and dispensed participants.
Arm/Group | Nelfilcon A | Etafilcon A
Serious Adverse Events (participants affected / at risk) | 2/234 | 0/235
Other Adverse Events (participants affected / at risk) | 0/234 | 0/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelfilcon A (N=234) | Etafilcon A (N=235)
Appendicitis (Surgical and medical procedures) | 1 (1) | 0 (0) — Unrelated
Foot injury requiring hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.